CLINICAL TRIAL: NCT01941888
Title: Phase IV Study of Propofol TCI (Target Controlled Infusion)Administered by Gastroenterologists During Endoscopy in Moderate Sedation: a Randomized Double Blind Controlled Study
Brief Title: Propofol TCI Administered by Gastroenterologists During Endoscopy: a Randomized Double Blind Controlled Study
Acronym: PropTCI/2012
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Agostoni Massimo, MD, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PropTCI2012
Record Dates: First submitted 2013-09-03; First posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Propofol; Target Controlled Infusion; Moderate Sedation; Gastrointestinal Endoscopy
MeSH Terms: interventions — Propofol; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol (Experimental): Patients in Group Propofol(n=70) were seated with propofol target concentration 1.2-1.6 µg/ml. Patients in both groups undergoing CS received also iv fentanyl (1μg/Kg) for pain control.
  Interventions: Drug: Propofol; Device: Target Controlled Infusion
- midazolam (Active Comparator): Control Group: patients in Group midazolam (n=70) were sedated with midazolam 0.04 mg/kg if aged< 70 - 0.03 mg/kg if aged> 70. Patients in both groups undergoing CS received also iv fentanyl (1μg/Kg) for pain control.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Propofol
  Arms: propofol
Drug: Midazolam
  Arms: midazolam
Device: Target Controlled Infusion
  Arms: propofol

SUMMARY:
Many studies address safety and effectiveness of non-anesthesiologist propofol sedation (NAPS) for GI endoscopy. Target Controlled Infusion (TCI) is a sophisticated tool for providing optimal sedation regimen and avoiding under or oversedation.

This randomized double blind controlled study compares standard moderate sedation level of sedation (group S) during upper endoscopy (EGD) and colonoscopy (CS) versus propofol NAPS (group P).

DETAILED DESCRIPTION:
70 CS and 70 EGD ASA I-II patients were studied. In group S (n=70) we administered fentanyl (1μg/kg) + midazolam (0.04-0.03 mg/kg) for CS and midazolam (0.04-0.03 mg/kg) for EGDS and in group P (n=70) fentanyl 1µg/Kg + propofol TCI 1.2-1.6 μg/ml for CS and propofol TCI 1.2-1.6 μg/ml for EGD. Vital parameters and Observer's Assessment of Alertness and Sedation Scale (OAA/S) were monitored throughout the study. Endoscopist's and patient's satisfactions were measured after procedure and 24-72 h later by visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* age >18 yrs
* ASA (American Society of Anesthesiologists risk class III-IV)I-II
* patients undergoing to gastroscopy or colonoscopy

Exclusion Criteria:

* significant systemic disease (American Society of Anesthesiologists risk class III-IV)
* history of allergic reactions to any of the study drugs
* chronic use of opioid analgesics
* psychiatric disorder
* pregnancy
* difficult airways (Mallampati score >2)
* age <18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Endoscopist's VAS (Visual Analog Scale) satisfaction about propofol TCI moderate sedation | one day
  Endoscopist's satisfaction was measured after endoscopic procedures by visual analog scale (VAS 0-100).
Patient's VAS (Visual Analog Scale) satisfactions about propofol TCI moderate sedation | one day
  Patient's satisfactions were measured after endoscopic procedures and 24-48 hours later by visual analog scale (VAS 0-100).

SECONDARY OUTCOMES:
Safety (number of partecipants with adverse events) of propofol TCI moderate sedation | one day
  To compare safety (number of partecipants with adverse events) of propofol TCI versus midazolam iv boluses during upper endoscopy (EGD) and colonoscopy (CS). Both sedation regimens were administered by endoscopists.
Time to dischargeability (minutes to reach Modified Aldrete score ≥ 18) of patients | one day
  To compare time to dischargeability (minutes to reach Modified Aldrete score ≥ 18) of patients in group standard versus propofol TCI group
  safety (number of partecipants with adverse events) of propofol TCI versus midazolam iv boluses during upper endoscopy (EGD) and colonoscopy (CS). Both sedation regimens were administered by endoscopists.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Agostoni, MD, Study Director — San Raffele Hospital; Lorella Fanti, MD, Principal Investigator — San Raffaele Hospital; Marco Gemma, MD, Principal Investigator — San Raffaele Hospital
Locations (2):
- Italy (2):
  - San Raffaele Hospital, Milan, Milan
  - San Raffaele Hospital, Milan